CLINICAL TRIAL: NCT00364949
Title: Genes, Androgens and Intrauterine Environment in PCOS
Brief Title: Intrauterine Environment in Polycystic Ovary Syndrome (PCOS) Probands
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Andrea Dunaif, Charles F Kettering Professor of Endocrinology & Metabolism Vice Chair for Research, Department of Medicine, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Other Study IDs: P50HD044405 (NIH)
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Results first posted 2010-08-18 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; PCOS; Pregnant; Cord Blood
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood

SUMMARY:
Polycystic ovary syndrome (PCOS) is among the most common endocrine disorders in premenopausal women, affecting 7-10% of this population. This syndrome is characterized by elevated levels of testosterone and chronic anovulation, and frequently of obesity. This study is designed to test the hypothesis that there is in utero testosterone excess, altered insulin secretion, and/or intrauterine growth retardation in the female offspring of women with PCOS. The allele 8 can be used to identify the reproductive and metabolic abnormalities associated with PCOS. This study will determine whether allele 8 positive [A8(+)] female offspring have more profound changes in these parameters compared to A8(-) female offspring.

Androgen and insulin levels in amniotic fluid from pregnant women with PCOS will be compared to levels in pregnant control women. Androgen and insulin levels in cord blood will also be measured. Further, gestational age and anthropomorphic measurements in offspring of women with PCOS will be assessed and compared to that in offspring of matched control women.

We will test the hypothesis that androgens are elevated in infancy in the female offspring of women with PCOS. We will assess sex steroids, insulin, and c-peptide levels in infants of PCOS women and compare them to the levels in infants of control women up to 1 year of age during the minipuberty of infancy. We will determine whether any of these parameters differ in A8(+) compared to A8(-) PCOS offspring.

DETAILED DESCRIPTION:
BACKGROUND Polycystic ovary syndrome (PCOS) is among the most common endocrine disorders in premenopausal women, affecting 7-10% of this population. This syndrome is characterized by hyperandrogenism, chronic anovulation and, frequently, obesity. Hyperandrogenemia seems to be a consistent reproductive phenotype in male relatives as well as female relatives of PCOS women. This phenotype appears to have a genetic basis in PCOS families and shows significant linkage and association with a marker locus on chromosome 19p in the region of the insulin receptor (allele 8 of D19S884.). This allele is also recently found to be associated with a metabolic phenotype in PCOS probands and their brothers, including increased post-challenge glucose levels, apparent defects in insulin secretion, especially in response to sulfonylurea, and accelerated weight gain with age (unpublished date). Therefore, allele 8 status in PCOS probands and their family members can identify the reproductive and metabolic abnormalities.

Many epidemiologic studies showed a plausible link between low birth weight and chronic metabolic disorders manifested as hypertension, diabetes and obesity later in life, suggestive of an early fetal programming. There is evidence to support fetal origin of PCOS. Female rhesus monkeys that were exposed to excess androgen in utero, were born smaller for gestational age. These animals had many of the reproductive features of PCOS, including increased LH levels, irregular ovulation, polycystic ovaries and functional ovarian hyperandrogenism. Similarly, in retrospective cohort studies, girls with elevated adrenal androgen levels or with PCOS were significantly smaller for gestational age at birth than reproductively normal control girls, suggestive of a possible fetal origin for some features of PCOS in human studies. Molecular mechanism for fetal programming is not clearly understood, but permanent changes in gene expression caused early insult may be a factor.

HYPOTHESIS These observations have led to a new hypothesis for the etiology of PCOS; genetic variation resulting in hyperandrogenemia leads to many of the reproductive and metabolic features of PCOS later in life. We will directly test the hypothesis that there is an excess androgen production in female offspring of women with PCOS. Further, we will test whether A8(+) female offspring have more profound changes in these parameters (increased androgen and/or decreased insulin levels in fetal life and in infancy) compared to A8(-) female offspring.

ELIGIBILITY:
Probands who meet the following criteria will be enrolled:

Menses < 6 per year without confounding meds Not taking confounding medications at the time of hormone analysis, willing to be off confounding medications for required washout period, or able to provide documentation of hyperandrogenemia (without hyperprolactinemia or evidence of non-classical adrenal hyperplasia) with past laboratory tests during a time when not taking confounding medications Total Testosterone >58 ng/dl or bioavailable testosterone >15 ng/dl Prolactin <25 ng/ml Baseline 17-OHP <3 ng/ml (and stimulated 17-OHP <10 ng/ml if subject is studied on-site)

Control women who meet the following criteria will be enrolled:

History of completely regular menstrual cycles. No history of hirsutism or alopecia. Control women will have a blood sample obtained 3-6 months after they have stopped lactating and resumed regular menses to ensure that they have normal T, uT and DHEAS levels.

Any pregnant woman who develops gestational diabetes will be excluded from the analysis.

To exclude disorders associated with insulin resistance, control subjects will have no personal history of hypertension or hypertriglyceridemia and no first-degree relative with Type 2 DM

Exclusion Criteria:

* history of gestational diabetes mellitus, eclampsia, pre-eclampsia or any medical disorders complicating their pregnancies.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women with PCOS and control women and their offspring
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2003-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea E Dunaif, MD, Principal Investigator — Chief, Division of Endocrinology, Metabolism and Molecular Medicine
Locations (1):
- Northwestern University School of Medicine, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: letters to participants from other studies and patients from Ob/Gyn at Northwestern
Pre-assignment Details: Exclusion based on personal/family history of diabetes or pre-existing medical condition
Groups:
- Control: Control
- PCOS: Polycystic Ovary Syndrome
Period: Overall Study
Arm/Group | Control | PCOS
Started | 31 | 39
Completed | 31 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | PCOS | Total
Number analyzed (Participants) | 31 | 39 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 39 | 70
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 39 | 70
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 39 | 70
Pre-pregnancy BMI [Mean (Standard Deviation); unit: kg/"m^2"] | 25.1 (5.7) | 30.8 (8.9) | 28.3 (7.5)
Maternal age at delivery [Mean (Standard Deviation); unit: yr] | 32.4 (4.4) | 30.1 (3.9) | 31.1 (4)

OUTCOME MEASURES:

1. Primary Outcome: Estradiol Level in Female Offspring
Description: The blood that were analyzed were taken from cord blood and not from the offspring.
Time Frame: One time sampling from the cord blood
Population: The number of the participants analyzed only included the levels for the female offspring.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | PCOS
Number analyzed (Participants) | 12 | 17
pg/ml | 18606 (18845) | 6467 (3989)
Statistical Analysis 1: Comparison: Control vs PCOS; Test type: Superiority or Other; p = 0.049, t-test, 2 sided

2. Primary Outcome: Androstenedione Level in Female Offspring
Time Frame: cord blood
Population: The number of participants analyzed only included the levels of the female offspring.
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Control | PCOS
Number analyzed (Participants) | 14 | 17
ng/dl | 146 (104) | 87 (46)
Statistical Analysis 1: Comparison: Control vs PCOS; Test type: Superiority or Other; p = 0.042, t-test, 2 sided

3. Primary Outcome: Testosterone Level in Female Offspring
Time Frame: cord blood
Population: The number of participants analyzed only included the levels of the female offspring.
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Control | PCOS
Number analyzed (Participants) | 14 | 16
ng/dl | 19 (29) | 7 (1)
Statistical Analysis 1: Comparison: Control vs PCOS; Test type: Superiority or Other; p = 0.156, t-test, 2 sided

4. Primary Outcome: 17-hydroxyprogesterone Level in Female Offspring
Time Frame: cord blood
Population: The number of participants analyzed only included the levels of the female offspring.
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Control | PCOS
Number analyzed (Participants) | 14 | 17
ng/dl | 2990 (1883) | 2777 (2103)
Statistical Analysis 1: Comparison: Control vs PCOS; Test type: Superiority or Other; p = 0.770, t-test, 2 sided

5. Primary Outcome: Dihydrotestosterone Level in Female Offspring
Time Frame: cord blood
Population: The number of participants analyzed only included the levels of the female offspring.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control | PCOS
Number analyzed (Participants) | 13 | 14
pg/ml | 88 (75) | 137 (162)
Statistical Analysis 1: Comparison: Control vs PCOS; Test type: Superiority or Other; p = 0.325, t-test, 2 sided

6. Primary Outcome: Dehydroepiandrosterone Level in Female Offspring
Time Frame: cord blood
Population: The number of participants analyzed only included the levels of the female offspring.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control | PCOS
Number analyzed (Participants) | 11 | 10
ng/ml | 5 (4) | 3 (2)

7. Primary Outcome: Infant Birth Weight (Male and Female)
Time Frame: birth
Population: Birth weight of the male and female infants.
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Control | PCOS
Number analyzed (Participants) | 31 | 39
gram | 3571 (389) | 3539 (597)

ADVERSE EVENTS:
Description: Serious and/or other (non-serious) adverse events were not assessed or collected because the cord blood sampling after the delivery of the offspring did not put anybody at risk.
Arm/Group | Control | PCOS
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/39
Other Adverse Events (participants affected / at risk) | 0/31 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No